CLINICAL TRIAL: NCT02209415
Title: Endoscopic Ultrasound (EUS) and PET-CT Based Follow-up of Patients Radically Resected for Cancer of the Oesophagus, Stomach or Pancreas.
Brief Title: EUFURO - EUS-based Follow-Up on R0-resected Patients for Esophageal, Gastric and Pancreatic Cancer
Acronym: EUFURO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michael Bau Mortensen (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Michael Bau Mortensen, MD, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-41-5702
Record Dates: First submitted 2011-11-28; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Esophageal Cancer; Stomach Cancer; Pancreatic Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard outpatient follow-up (Active Comparator): Outpatient clinic visits 3,6,9,12,18 and 24 mths after surgery
  Interventions: Behavioral: standard follow-up
- Intervention PET/CT and EUS (Experimental): PET/CT and EUS at 3,6,9,12,18 and 24 months after surgery
  Interventions: Procedure: PET/CT and EUS

INTERVENTIONS:
Behavioral: standard follow-up — Outpatient clinic visits
  Arms: Standard outpatient follow-up
Procedure: PET/CT and EUS — PET/CT and EUS
  Arms: Intervention PET/CT and EUS

SUMMARY:
Follow-up after successful operative treatment of cancer in the esophagus, stomach or pancreas in order to detect recurrent disease is a controversial topic.

This is because the methods and the consequence of following these patients is unknown.

Therefore the investigators will randomize these patients in to two groups:

1. One group of patients will be offered visits with a specialist surgeon in a outpatient setting for a clinical evaluation every 3,6,9,12,18 and 24 months after surgery, as is the current standard at our department.
2. The other group will be offered Endoscopic UltraSound, EUS, and PET/CT with the same intervals as the first group.

ELIGIBILITY:
Inclusion Criteria:

* R0- resection for primary adenocarcinoma or squamous cell carcinoma of the esophagus, stomach or pancreas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2011-04; Primary Completion 2016-01 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients eligible for treatment | 2 years
  Does early detection of recurrent disease translate in to more patients being eligible for oncologic treatment?

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Surgical Ultrasound, Department of upper surgical gastroenterology, Odense, Region Syddanmark, Denmark

REFERENCES:
- [Derived] Bjerring OS, Fristrup CW, Pfeiffer P, Lundell L, Mortensen MB. Phase II randomized clinical trial of endosonography and PET/CT versus clinical assessment only for follow-up after surgery for upper gastrointestinal cancer (EUFURO study). Br J Surg. 2019 Dec;106(13):1761-1768. doi: 10.1002/bjs.11290. Epub 2019 Oct 9. PMID 31595970
- [Derived] Bjerring OS, Hess S, Fristrup CW, Hoilund-Carlsen PF, Mortensen MB. The impact of endoscopic ultrasound-guided fine-needle aspiration of lymph nodes on subsequent positron emission tomography/computed tomography imaging: a prospective study. Endoscopy. 2019 Feb;51(2):165-168. doi: 10.1055/a-0647-6824. Epub 2018 Jul 23. PMID 30036892